CLINICAL TRIAL: NCT01942096
Title: Study of Airway Inflammation in Relation to Exercise in Elite Athletes
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dominque Bullens, prof dr, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: ML7650
Record Dates: First submitted 2013-08-26; First posted 2013-09-13 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Exercise Induced Asthma
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — induced sputum sample nasal fluid venous blood (serum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Competitive swimmers: Swimmers performing at national or international level
- Competitive indoor athletes: Indoor athletes performing at national or international level
- Healthy control individuals: Individuals performing sports at a recreational level

SUMMARY:
High school elite training programs are today more and more under development in several 'elite sport schools' in Belgium, in order to select and train future elite athletes already at young age. Little is known about the effects of sustained training on the potential development of asthma in adolescents during lung growth. It would be of great importance to be able to select the individuals at risk to develop exercise-induced asthma, already at the start of their enrollment in the 'elite sport school. This would allow physicians to follow their lung function parameters very closely and regularly; and, if necessary, start treatment early after the first signs of exercise-induced asthma.

DETAILED DESCRIPTION:
Competitive swimmers, competitive indoor athletes and control individuals performing sports at a recreational level will be recruited for the study.

They will perform a sport-specific training (swimmers and controls: swimming for 90 minutes, indoor athletes: basketball or volleyball for 90 minutes)

Baseline measurements:

* Airway inflammation upper and lower airways will be assessed by collection of nasal fluid (nasal sponge will be inserted in nostril for 5 minutes), Fraction of exhaled Nitric Oxide measurement and sputum induction.
* Upper and lower airway symptoms will be assessed by questionnaires (SinoNasal Outcome Measure-22, Visual Analogue Score, Asthma Symptom Score and Juniper Score)
* Allergy will be assessed by skin prick test (on skin) and immunocap test (in blood, 1 tube of 10 ml).
* Lung function and nasal patency will be measured by spirometry and Peak Nasal Inspiratory Flow measurement.
* Exercise induced bronchoconstriction will be assessed by eucapnic voluntary hyperventilation test.

Measurements immediately after training:

* Collection of nasal fluid
* Assessment of upper airway symptoms (Visual Analogue Score)
* Spirometry and Fraction of Exhaled Nitric Oxide measurement
* Peak Nasal Inspiratory Flow measurement

Measurements 24 hours after training:

* Collection of nasal fluid
* Assessment of upper airway symptoms (Visual Analogue Score)
* Spirometry and Fraction of Exhaled Nitric Oxide measurement
* Peak Nasal Inspiratory Flow measurement
* Sputum induction
* Venous puncture (1 tube of 10 ml)

ELIGIBILITY:
Inclusion Criteria:

* Performing sports at national or international level (swimmers and indoor athletes)

Exclusion Criteria:

* Performing sport at recreational level (not more than 4 hours/week for healthy individuals)

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Competitive swimmers, competitive indoor athletes and healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Measurement of airway inflammation | Baseline, immediately after and 24 hours after sport-specific training
  Airway inflammation upper and lower airways will be assessed by collection of nasal fluid (nasal sponge will be inserted in nostril for 5 minutes), Fraction of exhaled Nitric Oxide measurement and sputum induction.

SECONDARY OUTCOMES:
Measurement of exercise induced bronchoconstriction | baseline
  Exercise induced bronchoconstriction will be assessed by eucapnic voluntary hyperventilation test.

OTHER OUTCOMES:
Detection of allergy | baseline
  -Allergy will be assessed by skin prick test (on skin) and immunocap test (in blood, 1 tube of 10 ml).
Assessment of upper and lower airway symptoms | Baseline, immediately after and 24 hours after sport-specific training
  -Upper and lower airway symptoms will be assessed by questionnaires (SinoNasal Outcome Measure-22, Visual Analogue Score, Asthma Symptom Score and Juniper Score)
Measurement of lung function and nasal patency | at baseline, immediately after and 24 hours sport-specific training
  -Lung function and nasal patency will be measured by spirometry and Peak Nasal Inspiratory Flow measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Sven F Seys, MSc, Study Director — lab of clinical immunology, CDG 8th floor, Herestraat 49, 3000 Leuven; Valerie Hox, MD, Study Director — lab of clinical immunology, CDG 8th floor, Herestraat 49, 3000 Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Overall results are presented in a closed session for participants and parents. Confidential individual data are afterwards discussed with the respective parents and participants.

REFERENCES:
- [Result] Steelant B, Hox V, Van Gerven L, Dilissen E, Dekimpe E, Kasran A, Aertgeerts S, Van Belle V, Peers K, Dupont LJ, Hellings PW, Bullens DM, Seys SF. Nasal symptoms, epithelial injury and neurogenic inflammation in elite swimmers. Rhinology. 2018 Sep 1;56(3):279-287. doi: 10.4193/Rhin17.167. PMID 29561921
- [Result] Seys SF, Hox V, Van Gerven L, Dilissen E, Marijsse G, Peeters E, Dekimpe E, Kasran A, Aertgeerts S, Troosters T, Vanbelle V, Peers K, Ceuppens JL, Hellings PW, Dupont LJ, Bullens DM. Damage-associated molecular pattern and innate cytokine release in the airways of competitive swimmers. Allergy. 2015 Feb;70(2):187-94. doi: 10.1111/all.12540. PMID 25358760